CLINICAL TRIAL: NCT02007850
Title: Effect of Continuous Femoral Analgesia on Quadriceps Muscle Strength-0.2% Ropivacaine Continuous Infusion Versus Patient Controlled Femoral Analgesia
Brief Title: Effect of Mode of Femoral Nerve Analgesia on Quadriceps Muscle Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hae Wone Chang, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1308/214-010
Record Dates: First submitted 2013-10-28; First posted 2013-12-11 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Muscle Weakness
Keywords: continuous femoral nerve block; knee arthroplasty; quadriceps muscle strength
MeSH Terms: conditions — Muscle Weakness | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine continuous mode (Placebo Comparator): 0.2% ropivacaine 8 ml/hr through femoral nerve block catheter for 2 days and they have patient controlled intravenous fentanyl
  Interventions: Drug: ropivacaine
- ropivacaine patient controlled mode (Active Comparator): 0.2% ropivacaine patient controlled mode, basal rate 4 ml/hr, bolus 4 ml, lockout 60 minutes through femoral nerve block catheter for 2 days and they have patient controlled intravenous fentanyl
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — Patients receive 15 ml of 0.25% ropivacaine pre-operatively through femoral block catheter, followed by 0.2% ropivacaine continuous mode or patient controlled mode for 2 days after surgery
  Other Names: femoral nerve block

SUMMARY:
Quadriceps muscle strength is an important determinant of quality of recovery in elderly patients after total knee arthroplasty. We try to compare the quadriceps muscle strength change between 0.2 % ropivacaine continuous fixed femoral infusion and patient controlled femoral analgesia group.

DETAILED DESCRIPTION:
Continuous femoral nerve analgesia technique is relatively safe, can be easily trained, and reduces significantly intravenous opioid consumption. These favorable features make it standard treatment option for postoperative knee pain. However, direct perineural local anesthetic effect is not only confined into pain fiber, but, the other sensory and motor nerve fibers. Therefore, unwanted motor weakness is accompanied. Quadriceps muscle strength, which is important determinant of physical function after knee arthroplasty, can be influenced in continuous femoral nerve block. Various local anesthetic infusion techniques have been suggested to minimize the change of quadriceps muscle strength. Decreasing local anesthetic concentrations affect not only degree of muscle weakness, but also reduces the quality of pain control. Different anatomic location of catheter tip, considering motor fiber in posterior part of femoral nerve, could not reduce motor weakness. In a study with continuous popliteal-sciatic nerve blocks after hallux valgus repair, repeated bolus administration seems to be more effective method for pain control without concurrent motor impairment. However, another study with continuous femoral nerve block in healthy volunteers, hourly repeated bolus dose of 5 ml of 0.1% ropivacaine failed to spare motor block. Previously, our institution standard technique is fixed continuous infusion of 0.2% ropivacaine and concomitant intravenous patient controlled fentanyl. Because physical therapy of our institution, usually starts with the 2nd day of operation, so, we assume that continuous fixed infusion may result in more drug accumulation near nerve fiber. So, patient controlled mode of femoral analgesia could be better choice for initiation of physical therapy. At the same time, comparison between patient controlled analgesia and continuous infusion is not fully elucidated until recently. Therefore, in this study, we try to compare quadriceps muscle strength change between continuous infusion and patient controlled femoral analgesia in patients undergoing total knee replacement arthroplasty. Secondary outcomes include sensory effect in femoral nerve distribution, pain scores, iv fentanyl consumption, and other adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* > 21, or < 80 years old- men and women
* primary, unilateral total knee replacement surgery
* spinal anesthesia

Exclusion Criteria:

* general anesthesia
* secondary knee replacement surgery
* patient refusal for continuous femoral nerve analgesia technique
* abnormal coagulation profile, e.g. Prothrombin time international normalized ratio > 1.5, activated partial thrombin time > 50 sec
* within 5 days after termination oral antiplatelet agent
* Body mass index>45
* impaired renal function
* infection near femoral area
* previous injury near femoral area
* neurologic dysfunction in lower limb
* previous adverse drug reaction for local anesthetics
* American society of anesthesiologists (ASA) class III, iV or V

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change of quadriceps muscle strength | Baseline, Postoperative 2nd day
  maximum voluntary isometric contraction of quadriceps femoris with hand held manometry

SECONDARY OUTCOMES:
sensory changes in femoral nerve distribution | postoperative 2 day
  tolerance to transcutaneous electrical stimulation
pain scores | postoperative 1 day
  verbal numeric pain scale (0-100) resting/dynamic
pain scores | postoperative 2 day
  verbal numeric pain scale (0-100) resting/dynamic
intravenous fentanyl consumption | postoperative 2 day
  cumulative fentanyl consumption on postoperative 2 day

CONTACTS AND LOCATIONS:
Overall Officials: Hae Wone Chang, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Sungnam, Gyungido, South Korea